CLINICAL TRIAL: NCT07296471
Title: An Observational Study to Explore the Associations Between Vitamin D Status and Genomic, Proteomic, and Metabolomic Profiles in Patients With Primary Osteoporosis
Brief Title: Vitamin D Status and Multi-Omics Profiles in Primary Osteoporosis
Acronym: OP-MultiOmics
Status: Recruiting | Type: Observational
Sponsor: Dr. Li Chen (Other)
Responsible Party: Sponsor-Investigator, Dr. Li Chen, Associate Chief Physician, Department of Laboratory Medicine, Yichang Second People's Hospital, Yichang Second People's Hospital
Organization: Yichang Second People's Hospital (Other)
Other Study IDs: YCSR202526
Record Dates: First submitted 2025-11-14; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Primary Osteoporosis
Keywords: Primary Osteoporosis; Vitamin D; Multi-omics; Transcriptomics; Proteomics; Metabolomics; Biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Osteoporosis Patients: Adults newly diagnosed with primary osteoporosis (n=90) at Yichang Second People's Hospital. Blood and serum samples will be collected at the initial visit for transcriptomic, proteomic, and metabolomic analyses. No additional research sampling or follow-up will be performed.
- Healthy Controls: Healthy adults without osteoporosis (n=30) at Yichang Second People's Hospital. Blood and serum samples will be collected at the initial visit for transcriptomic, proteomic, and metabolomic analyses. No additional research sampling or follow-up will be performed.

SUMMARY:
This observational study aims to explore the relationships between vitamin D status and genomic, proteomic, and metabolomic profiles in patients with primary osteoporosis.

Eligible participants are adults who are newly diagnosed with primary osteoporosis at Yichang Second People's Hospital. Blood samples will be collected at the initial diagnosis to analyze gene expression, protein levels, and metabolic profiles.

Participants will receive standard clinical treatment according to routine care, but no additional research sampling or follow-up will be performed.

The study seeks to identify molecular patterns associated with osteoporosis and improve understanding of patient responses to therapy.

DETAILED DESCRIPTION:
This observational study will enroll adults newly diagnosed with primary osteoporosis at Yichang Second People's Hospital.

Blood samples will be collected at the initial diagnosis for multi-omics analysis, including transcriptomics, proteomics, and metabolomics. Clinical data, including bone mineral density, serum calcium, and vitamin D levels, will also be collected.

No additional research sampling or follow-up is planned after the initial visit.

Data analysis will focus on identifying molecular patterns associated with osteoporosis and potential biomarkers related to vitamin D status. All procedures will follow ethical guidelines and standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy controls: Adults aged ≥18 years, with normal bone mineral density (BMD) confirmed by dual-energy X-ray absorptiometry (DXA), without a history of bone metabolic diseases, major organ dysfunction, or chronic inflammatory/autoimmune diseases.
2. Osteoporotic patients: Adults aged ≥18 years, newly diagnosed with primary osteoporosis according to clinical criteria (T-score ≤ -2.5 SD by DXA), without serious complications that may affect study results.
3. Participants willing and able to provide written informed consent and cooperate with study procedures, including blood and serum sample collection and clinical data recording.

Exclusion Criteria:

1. Patients with secondary osteoporosis, including but not limited to osteoporosis caused by hyperparathyroidism, tumors, chronic kidney disease, liver cirrhosis, rheumatoid arthritis, or other autoimmune diseases.
2. Individuals who have taken vitamin D supplements, anti-osteoporotic drugs, glucocorticoids, or other medications affecting vitamin D or bone metabolism within 3 months prior to enrollment.
3. Pregnant or lactating women, or individuals with mental disorders preventing cooperation with study procedures.
4. Individuals with acute infections, malignant tumors, or severe liver, kidney, cardiovascular, or cerebrovascular diseases that may affect study outcomes.
5. Participants with a history of blood transfusion within 1 month prior to enrollment or those unable to provide peripheral blood samples as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the outpatient and inpatient population of Yichang Second People's Hospital, including adults newly diagnosed with primary osteoporosis as well as healthy adult volunteers. Blood and serum samples will be collected at the hospital laboratory for multi-omics analyses.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Gene Expression Profiles Derived From Transcriptomic Analysis | Baseline
  Quantitative gene expression levels obtained from whole blood RNA sequencing, including the identification of differentially expressed genes and their expression magnitudes (e.g., log2 fold change, normalized counts).
Serum Protein Abundance Profiles From Proteomic Analysis | Baseline
  Quantitative abundance of serum proteins measured through mass spectrometry-based proteomics, including identification of differentially expressed proteins and their relative abundance levels.
Serum Metabolite Abundance Profiles From Metabolomics Analysis | Baseline
  Quantitative serum metabolite abundance determined by untargeted metabolomics, including identification of metabolites with altered abundance and their relative intensity values.

SECONDARY OUTCOMES:
Bone Mineral Density (BMD) | Baseline
  Bone mineral density measured at the lumbar spine and/or hip using dual-energy X-ray absorptiometry (DXA).
Serum 25-Hydroxyvitamin D Level | Baseline
  Serum concentration of 25-hydroxyvitamin D (25(OH)D) assessed at enrollment to evaluate vitamin D status.
Serum Calcium Level | Baseline
  Serum calcium concentration measured at enrollment as a routine biochemical indicator of bone metabolism.
Serum Phosphate Level | Baseline
  Serum phosphate concentration measured at enrollment to assess mineral metabolism status.
Serum Magnesium Level | Baseline
  Serum magnesium concentration measured at enrollment as part of biochemical evaluation related to bone health.
Serum Osteocalcin Level | Baseline
  Serum osteocalcin concentration measured as a marker of bone formation.
Serum Alkaline Phosphatase (ALP) | Baseline
  Serum alkaline phosphatase level assessed as an indicator of bone turnover and metabolic activity.
Serum β-CTX Level | Baseline
  Serum C-terminal telopeptide of type I collagen (β-CTX) measured to evaluate bone resorption activity.
Serum P1NP Level | Baseline
  Serum procollagen type 1 N-terminal propeptide (P1NP) measured as an additional bone formation marker.

CONTACTS AND LOCATIONS:
Locations (1):
- Yichang Second People's Hospital, Yichang, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including multi-omics datasets (transcriptomic, proteomic, metabolomic) and clinical measurements will be shared with qualified researchers upon reasonable request.
Supporting Information: Study Protocol
Time Frame: De-identified individual participant data and supporting information will be available to qualified researchers starting after publication of the primary study results and will remain available for at least 5 years.
Access Criteria: De-identified individual participant data and supporting information will be accessible to qualified researchers who submit a reasonable proposal and agree to a data use agreement. Data will be shared electronically after approval of the request.